CLINICAL TRIAL: NCT04502173
Title: Kenya: An Implementation Study on the Barriers and Facilitators of Scaling up the Innovative, Low-cost Ellavi Uterine Balloon Tamponade for Postpartum Hemorrhage
Brief Title: Kenya: The Barriers and Facilitators of Scaling up the Ellavi UBT for Postpartum Hemorrhage
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Collaborators: Department for International Development, United Kingdom (Other Government); University of Nairobi (Other)
Responsible Party: Principal Investigator, Megan Parker, Principal Investigator, PATH
Other Study IDs: 1512602-2
Record Dates: First submitted 2020-06-11; First posted 2020-08-06 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training: Study participants trained on how to use the Ellavi intra-uterine balloon tamponade via virtual webinar training. Feedback on training course elements will be obtained for future improvements prior to scaling.
  Interventions: Device: Ellavi UBT
- Managing PPH: Study participants who provided refractory PPH care using an Ellavi UBT device will give feedback on the barriers and facilitators to use of the newly registered, low-cost medical device.
  Interventions: Device: Ellavi UBT

INTERVENTIONS:
Device: Ellavi UBT — The study team will train all obstetric healthcare staff (i.e. obstetricians, midwives, medical officers, clinical officers) involved in PPH management at the participating healthcare facilities on use of the Ellavi UBT. This will be done to gather feedback from the healthcare workers (post-training and post-PPH) to understand the barriers to and facilitators of use in order to evaluate acceptability and feasibility among facilities providing different levels of care (level 4, level 5 (county), level 6 (tertiary)).

SUMMARY:
The purpose of this implementation research study is to generate evidence that informs the successful uptake and adoption of the Ellavi Uterine Balloon Tamponade (UBT) within Kenyan postpartum hemorrhage (PPH) management programs. The investigators aim to improve the likelihood that the Ellavi UBT will be integrated into the Kenyan health care system by obtaining critical feedback from stakeholders and health care providers on the barriers and facilitators towards its successful adoption and roll out. The research will be done in three purposively selected University of Nairobi affiliated hospitals in Nairobi county, Kenya. This study will therefore be exploratory and use a non-experimental design. The study team will train all obstetric healthcare staff (i.e. obstetricians, midwives, medical officers, clinical officers) involved in PPH management at the participating healthcare facilities on use of the Ellavi UBT. The investigators will then gather feedback from the obstetric healthcare workers (post-training and post-PPH) to understand the barriers to and facilitators of use in order to evaluate acceptability and feasibility among facilities providing different levels of care (level 4, level 5 (county), level 6 (tertiary)). This process will help to generate training and facility level recommendations for improved uptake and integration into the local maternal care package. Case report forms and semi-quantitative surveys will be completed by obstetrical care providers to evaluate the primary outcomes of acceptability and feasibility by measuring: context of use, accuracy of use, perceptions of the device, user confidence, acceptability, usability, facilitators of use, barriers to use, use-patterns, and insights into training effectiveness. The secondary outcomes will include financial data to determine the cost of introducing the Ellavi UBT into the Kenyan PPH management protocols and the health system. The study will not involve the storage of biological samples. There is not a direct benefit of the study to the individual participants. All study participants will sign consent forms.

DETAILED DESCRIPTION:
The purpose of this implementation research study is to generate evidence that informs the successful uptake and adoption of the Ellavi UBT within Kenyan MOH PPH management programs for both public and private sector programs. The investigators aim to generate evidence for Kenyan stakeholders to use in their decision-making around the use of Ellavi UBT in Kenyan PPH management programs.

Specific objectives:

1. To determine the adoption, penetration, sustainability and fidelity of implementing the Ellavi UBT device into PPH care in three health care facilities (2 public facilities, 1 private facility). The investigators will explore the number of health workers and facilities that receive the PPH and Ellavi UBT training, and percent of health workers and facilities that adopt the Ellavi UBT device over the 6-month period. The investigators will also assess factors that influence the adoption, penetration, sustainability, and fidelity through an operations research survey, and the Ellavi UBT questionnaire.
2. To determine the appropriateness, acceptability and feasibility of using the Ellavi UBT in participating health facilities at various levels of care in Nairobi County, the investigators will explore user comprehension of the Ellavi UBT usage steps, accuracy of use, perceptions of the device, attitudes towards the device, user confidence, usability, facilitators of use, barriers to use, use-patterns, and insights into training effectiveness.

   1. Sensitize senior management at each of the three participating facilities, separately.
   2. Conduct two half-day trainings on PPH and Ellavi UBT use at each of the three participating health facilities separated by: 1) obstetricians, medical and clinical officers, and 2) midwives.
   3. Collect individual initial (post-training) data to assess comprehension of Ellavi UBT usage steps, perceptions of the device, attitudes towards the device, user confidence, usability, and insights into training effectiveness.
   4. Case Management Form (CMF): Obstetrical care provider will complete a CMF within 24hrs (<24hrs) of managing each PPH event. This will inform the study team of how decision-making algorithms were applied and accuracy of use.
   5. Ellavi UBT Questionnaire: PATH-Kenya study team member will collect individual post (post-usage) Ellavi UBT use data (<72hrs) from each study participant (obstetrical care worker) to assess comprehension of Ellavi UBT usage steps, perceptions of the device, attitudes towards the device, user confidence, usability, facilitators of use, barriers to use, use-patterns, and insights into training effectiveness.
   6. PATH-Kenya study staff will record secondary data from hospital registry books over the six (6) month duration of this study (March - August 2020) in comparison to the same six (6) month period in 2019 to examine changes in use of condom catheters, and Ellavi UBTs.
   7. Use the Consolidated Framework for Implementation Research (CFIR) to identify constructs with the potential to influence the introduction and use of Ellavi UBT. These constructs will be mapped to questions in the questionnaire, and will be analyzed to identify their influence on Ellavi UBT use. Constructs that have influence on the implementation of UBTs (both positively and negatively) will be disseminated for use in future introduction and scale up of Ellavi UBTs.
3. To determine the cost of introducing the Ellavi UBT into the PPH management protocol and health system.

   1. Estimate the costs of the different obstetrical care provider training components.
   2. Estimate the costs for other country-level activities associated with the introduction of the UBT into the PPH management protocols such as costs for meetings, advocacy, and communication materials.
   3. Qualitatively evaluate the frequency and duration of stock outs of condoms, catheters, IV fluids (sterilized materials), and sutures.
   4. Estimate the costs of staff time spent on assembling a condom catheter UBT and the costs of supplies used.
4. To disseminate the information in national (KOGS), regional (ECSACOG, AFOG), and international forums to support information sharing, increased awareness of the role of UBT for refractory PPH, and adoption of its use.

   e. Summarize how the Ellavi UBT can be integrated into curriculums, guidelines, and hospital systems (e.g. patient-provider friendly materials) by analyzing the key facilitators and barriers.

   f. Host a national level meeting with Kenyan MOH stakeholders and participating facilities g. Publish and disseminate findings in a peer-reviewed journal h. Present at international conferences and forums, as funding permits. Show the use of Ellavi UBT using poster presentations and demonstration sessions at international obstetrics meetings: FIGO, WHO UBT group, Women Deliver as funding permits.

ELIGIBILITY:
Inclusion Criteria:

* Obstetricians, medical officers, clinical officers, and midwives who recently participated in a PPH/Ellavi UBT training or managed a refractory PPH case (with or without the use of an Ellavi UBT (within the past 72 hours) at one of the 3 participating health care facilities.
* Hospital administrators, supply store managers and/or procurement staff

Exclusion Criteria:

- Obstetricians, medical officers, clinical officers, and midwives working at the facility who do not agree or consent to participate.

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Obstetrical care providers who recently participated in a training (before using the Ellavi UBT device for case management) and/or obstetrical care providers who recently managed a refractory PPH event. The study participant must work in one of the three participating health care facilities. The number of interviewees per site will vary depending on the size of the facility and the number of refractory PPH events.
  Eligible participants will be selected based on their participation in a PPH/Ellavi UBT training session, or their management of a PPH event. The study participants will include obstetricians, midwives, medical officers and clinical officers currently practicing medicine at Kenyatta National Hospital, Mbagathi Hospital, or St. Mary's Mission Hospital. If a facility has only three obstetrical care providers, these people will be re-sampled for each refractory PPH event to understand their interactions with the Ellavi UBT each time.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Determine the appropriateness, acceptability and feasibility of using the Ellavi UBT via semi-quantitative surveys (quantitative and qualitative measures) with health care providers in Nairobi County. | 6 months
  Determine feasibility by measuring: 1) user comprehension of the Ellavi UBT usage steps and accuracy of use by evaluating assembly, timing of use, relevance for patient's health status (semi-quantitative measures), 2) facilitators of use and barriers to use (open ended, qualitative questions on facility placement, leadership influence, procurement channels, patient feedback), and 3) insights into training effectiveness (opened ended qualitative questions on preferred methods of training, quality of teaching provided). These outcome measures will be evaluated using both quantitative (multiple choice, likert scale) and qualitative (open ended explanations) responses.
  Determine acceptability by measuring: perceptions of the device (likert scale), attitudes towards the device (likert scale), user confidence (likert scale), and usability (likert scale).
  Determine appropriateness by measuring: patterns of use with open ended qualitative questions.
Determine the adoption, penetration, sustainability and fidelity of implementing the Ellavi UBT by examining hospital record books and collecting quantitative data. | 6 months
  Determine the adoption, penetration, sustainability and fidelity of implementing the Ellavi UBT device into PPH care at 3 health care facilities using semi-quantitative surveys and hospital level record books.
  Determine penetration: # facilities participating, # health workers trained, % of all health workers trained at each site.
  Determine adoption: % of facilities that adopted UBT devices, # of trained health workers who used the UBT.
  Determine sustainability: proportion of facilities and health worker who use UBTs/month, for 6 months; %l of providers that use the UBT correctly for >80% of cases.
  Determine fidelity: % of all health workers surveyed that used the Ellavi UBT.

SECONDARY OUTCOMES:
Determine the cost of introducing the Ellavi UBT into the PPH management protocol and health system by examining cost data, hospital procurement records, and quantifying labor hours worked. | 6 months
  Determine the costs of the different training course components by reviewing charges incurred.
  Determine the costs for country-level activities associated with UBT introduction into the PPH management protocols. This includes costs for meetings, advocacy, and communication materials (e.g. review spreadsheets of costs incurred).
  Determine the frequency and duration of stock outs of: condoms, catheters, IV fluids (sterilized materials), and sutures by surveying hospital inventory stock.
  Determine the costs of staff time spent on assembling a condom catheter UBT. Determine the costs of supplied pieces to assemble condoms catheters.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Parker, PhD, Principal Investigator — PATH
Locations (1):
- Kenyatta National Hospital, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No
The de-identified data will be shared with the funder in the form of a study report. If data are held on a public database (due to publication requirements), they will not be linked to the study participant and their identity would not be revealed.

REFERENCES:
- [Derived] Parker ME, Qureshi Z, Deganus S, Soki J, Cofie P, Dapaah P, Owusu R, Gwako G, Osoti A, Ogutu O, Opira J, Sunkwa-Mills G, Boamah M, Srofenyoh E, Aboagye P, Fofie C, Kaliti S, Morozoff C, Secor A, Metzler M, Abu-Haydar E. Introduction of the Ellavi uterine balloon tamponade into the Kenyan and Ghanaian maternal healthcare package for improved postpartum haemorrhage management: an implementation research study. BMJ Open. 2023 Feb 3;13(2):e066907. doi: 10.1136/bmjopen-2022-066907. PMID 36737079